CLINICAL TRIAL: NCT00361166
Title: A Randomized, Double Blind, Multi-Center Study to Assess the Antipsychotic and Motor Effects of ACP-103 When Administered in Combination With Haloperidol or Risperidone to Schizophrenic Subjects
Brief Title: Antipsychotic and Motor Effects of ACP-103 When Administered in Combination With Haloperidol and Risperidone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ACP-103-008
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2007-03-22 (Estimated); Status verified 2007-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; psychosis; delusions; hallucination
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Delusions; Hallucinations | interventions — pimavanserin

INTERVENTIONS:
Drug: ACP-103

SUMMARY:
The primary purpose of this study is to determine whether a combination of ACP-103 (the study medication) with either haloperidol or risperidone will show antipsychotic efficacy and that it is safe and well tolerated. Further purposes of this study are to determine whether ACP-103, in combination with either haloperidol or risperidone, will enhance their antipsychotic effectiveness, demonstrate effectiveness against the negative symptoms, improve motoric tolerability, and is safe and well tolerated.

This is a seven-week study (one week screening and six weeks of study medication) where a total of 400 patients who meet entrance criteria will randomly be assigned to receive one of five groups of study treatments of either low dose haloperidol plus ACP-103, low dose haloperidol plus placebo (a substance similar to a sugar pill), low dose risperidone plus ACP-103, low dose risperidone plus placebo, or high dose risperidone plus placebo. The study will begin with with a three to seven day drug-free period followed by six weeks of a stable daily dosage of study medication. Study subjects will be treated as hospital in-patients during screening and for the first 14 days of the study. Study subjects will be closely monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects ages 18-65 diagnosed with schizophrenia
* experiencing an acute exacerbation of psychosis
* has had prior response to antipsychotic therapy within the previous 3 years
* female subjects must be of non-childbearing potential or must comply with double-barrier protection methods against conception
* ability of subject or caregiver or legally authorized representative to provide informed consent
* subjects must be hospitalized at screening and must be willing to remain in the hospital at least 14 days after baseline and must comply with all study events through completion of the study

Exclusion Criteria:

* inability of the subject or caregiver or legally authorized representative to provide consent
* any female subject who is pregnant or breast feeding
* any subject with concurrent mental illness or disability
* any subject considered to be a danger to themselves or others
* recent use of certain antipsychotics or other medications that might interfere with this study's medication
* abnormal clinical laboratory values
* presence, or recent history, of serious medical conditions or drug abuse
* likely allergy or sensitivity to ACP-103, haloperidol, or risperidone, based on known allergies to drugs of the same class
* any subject who has participated in a prior clinical trial of ACP-103
* any subject judged by the Principal Investigator to be inappropriate for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Total score on the Positive and Negative Symptom Scale (PANSS).

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S), Simpson Angus Scale (SAS), Barnes Akathisia Scale (BAS), Calgary Depression Scale for Schizophrenia (CDSS)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel van Kammen, MD, PhD, Study Chair — ACADIA Pharmaceuticals Inc.
Locations (15):
- United States (10):
  - Cerritos, California
  - Garden Grove, California
  - Glendale, California
  - Paramount, California
  - Pico Rivera, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - St Louis, Missouri
  - Austin, Texas
  - Irving, Texas
- Brazil (5):
  - Salvador, Estado de Bahia
  - Aparecida de Goiânia, Goiás
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - São Paulo, São Paulo